CLINICAL TRIAL: NCT06791213
Title: Effectiveness of the Digital Multimedia Health Education in Improving Cancer Pain, Analgesic Adherence, and Pain Control Satisfaction With Cancer Patient
Acronym: EDICAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202407158RINE
Record Dates: First submitted 2025-01-13; First posted 2025-01-24 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-10

CONDITIONS: Cancer Pain
Keywords: Cancer Pain; Digital Multimedia Health Education; Analgesic Adherence; Pain Control Satisfaction
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Digital Multimedia Health Education
  Interventions: Other: Digital Multimedia Health Education
- Control group (No Intervention)

INTERVENTIONS:
Other: Digital Multimedia Health Education — This study aims to investigate the effectiveness of "digital multimedia" in reducing pain, enhancing medication adherence, and improving pain control satisfaction among patients. The goal is to overcome the limitations of busy healthcare providers, allowing patients to learn independently, understand pain and analgesic use, dispel myths about pain medications, and enhance pain control, ultimately improving self-care capabilities, pain control satisfaction, and quality of life.
  Arms: Treatment group

SUMMARY:
According to the International Association for the Study of Pain (IASP), pain is an unpleasant sensory and emotional experience associated with, or resembling that associated with, actual or potential tissue damage . Despite advances in precision medicine, pain remains a common complaint among cancer patients, with 44.5% reporting pain and a 30.6% prevalence of moderate to severe pain. In Taiwan, over half of cancer patients experience pain in the week leading up to their outpatient visit, with 54% of oncology outpatients reporting pain issues. Of these, only 58% receive analgesics, with more medications given to those with worsening conditions. Pain significantly affects sleep, and over 50% of patients feel pain despite analgesic control. Research indicates that Asian patients often view cancer negatively, avoiding discussions about their condition, which normalizes their pain and potentially worsens it.

Enhancing patient self-efficacy can increase satisfaction with pain management, and it is recommended that healthcare professionals develop interventions to improve pain management satisfaction. Self-management interventions have shown effectiveness in improving pain-related knowledge and quality of life. These interventions can encompass patient attitudes and knowledge, with guidance and consultation from nurses reinforcing information about pain management and medication adherence.

In clinical settings, nurses may be too busy to provide comprehensive and consistent health education, leading to insufficient patient understanding of medications. Digital multimedia health education tools, which use visual aids, can better capture patients' attention and facilitate unrestricted learning regardless of time or place, leading to improved learning outcomes.

This study aims to investigate the effectiveness of "digital multimedia" in reducing pain, enhancing medication adherence, and improving pain control satisfaction among patients. The goal is to overcome the limitations of busy healthcare providers, allowing patients to learn independently, understand pain and analgesic use, dispel myths about pain medications, and enhance pain control, ultimately improving self-care capabilities, pain control satisfaction, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18 years.
* Diagnosed with a solid tumor and reporting a pain score of 4 or higher.
* Patients using prescribed strong opioid medications for pain management.
* Conscious, capable of communicating in Mandarin, understanding Mandarin, or -Able to write in text.
* Able to operate electronic devices (e.g., smartphones, tablets, or computers) independently, or with assistance from family members or caregivers.

Exclusion Criteria:

* Patients with visual or auditory impairments.
* Patients with cognitive impairments.
* Diagnosed by a physician as having substance addiction (addictive substances include central nervous system depressants: opioids, heroin, ketamine; central nervous system stimulants: amphetamines, ecstasy, cocaine; and central nervous system hallucinogens: cannabis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Cancer pain | From enrollment to the end of treatment at 12 weeks
  This study defines its operational terms using the Taiwanese version of the Brief Pain Inventory (BPI-T). Pain is assessed through the Numerical Rating Scale (NRS), which evaluates pain severity on a scale ranging from 0 to 10. Higher scores indic.
Analgesic Adherence | From enrollment to the end of treatment at 12 weeks
  1. Calculate the total amount of pain medication consumed by patients and the total amount prescribed by physicians to determine the medication adherence percentage. Additionally, convert opioid prescriptions into morphine-equivalent doses to calculate the medication adherence percentage.
  2. The 4-item Morisky Medication Adherence Scale (MMAS-4) was used for assessment. This structured measurement scale was originally developed by Morisky et al. (1986) and consists of four questions. The MMAS-4 scores indicate medication adherence, with higher scores representing greater adherence to prescribed medication.
Pain Control Satisfaction | From enrollment to the end of treatment at 12 weeks
  The Pain Treatment Satisfaction Scale (PTSS) was adopted for psychometric assessment and validation in patients with acute and chronic pain. The scale evaluates various aspects, including pain severity, information about pain and its treatment, medication therapy, the effects of current pain medications, the route of administration, medication side effects, and satisfaction with current pain medications and overall care.

CONTACTS AND LOCATIONS:
Locations (1):
- 13F., No. 119, Ln. 136, Sec. 3, Zhongshan Rd., Zhonghe Dist., New Taipei City 235 , Taiwan (R.O.C.), New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No